CLINICAL TRIAL: NCT04751318
Title: Bioavailability of a Formulation of Duloxetine 60 mg Enteric Coated Granules With Regards to Reference Product in Feeding Conditions
Brief Title: Bioavailability of Duloxetine 60 mg With Regards to Reference Product in Feeding Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Andromaco S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP8825-01
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-02

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Duloxetine Hydrochloride; Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duloxetine Test Produc (Experimental): Participants will receive one capsule of the test formulation containing Duloxetine 60 mg. The capsules will be taken with water and in a feeding condition.
  Interventions: Drug: Duloxetine 60mg Test Drug Enteric Coated Granules
- Duloxetine Referent Product (Active Comparator): Participants will receive one capsule of the marketed reference formulation containing Duloxetine 60 mg. The capsules will be taken with water and in a feeding condition.
  Interventions: Drug: Duloxetine 60mg Reference Product Enteric Coated Granules

INTERVENTIONS:
Drug: Duloxetine 60mg Test Drug Enteric Coated Granules — Investigational Medicinal Product
  Other Names: Test Drug
  Arms: Duloxetine Test Produc
Drug: Duloxetine 60mg Reference Product Enteric Coated Granules — Cymbalta (Eli Lilly)
  Other Names: Reference Product
  Arms: Duloxetine Referent Product

SUMMARY:
This Study will investigate the bioavailability in fasting subjects of 1 capsule formulation containing Duloxetine 60 mg. The Study will be performed at a single site with 36 subjects.Participants will take 1 capsule of the test product and reference product in 2 periods and 2 sequences (either test after reference or reference after test). There will be a washout of at least 14 days between each study period.

DETAILED DESCRIPTION:
The primary objective of the study is to investigate the relative bioavailability of Duloxetine of 1 capsule formulation with Duloxetine 60 mg under feeding conditions to demonstrate bioequivalence of both formulations in terms of rate and extent of absorption:

* Test Product: Product manufactured by Laboratorios Andrómaco S.A.
* Reference Product: Cymbalta[Trademark], product of Eli Lilly, Puerto Rico.

The 90% confidence intervals for the intra-subject coefficient of variation (Test versus Reference Product) for the main pharmacokinetic parameters area under the plasma concentrationtime curve from time zero to time t (AUC0-t) and from time zero to 72 hours (AUC0-72), and maximum plasma concentration (Cmax) for total Duloxetine will be determined.

Participants will be confined in the study site for approximately 25,5 hours during each study period (for 10 hours pre-dosing and for 15,5 hours post dosing) during which pharmacokinetic (PK) blood samples will be obtained. 17 blood samples will be taken up to 24 hours after the administration in each period. Participants will return to the site to provide additional blood samples at 48 h, and 72 h postdose.The washout period between the two study periods will be at least 14 days.

The samples from each participant will be analyzed with 2 methods of high performance liquid chromatography-tandem mass spectrometry bioanalytical assays to quantify total Duloxetine in plasma.

The safety objective is to evaluate the tolerability of both formulations in subjects by collecting adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-breastfeeding women
* Women of childbearing age with an acceptable form of contraception during the study
* 18 to 55 years old inclusive; BMI greater than or equal to 18.51 and less than or equal to 29.99
* With results of laboratory tests, electrocardiogram and chest radiography in normal and / or negative or abnormal ranges but without clinical relevance and declared suitable for study by the doctor after the physical examination
* Capable to understand the Informed Consent Form

Exclusion Criteria:

* Study site staff or family members
* With history of drug and/or alcohol abuse
* Smokers more tan 3 cigarettes every 7 days
* Vitamin supplements intake 7 days prior to the administration of the medications under study
* Any recent change in eating habits or physical exercise
* Using of a pharmacological therapy (except over the counter medication use 7 days prior to the study)
* Hypersensitivity to the study drug or to other chemically related compounds, history of serious adverse reactions or hypersensitivity to any medication
* Use, during the 28 days prior to the start of the study, of medications known to alter liver enzyme activity
* Consumption of beverages or food containing grapefruit or pink grapefruit, within 7 days prior to each administration of the study medication and consumption of alcohol, caffeine or beverages or foods containing xanthines 24 hours before each administration of the study medication until the last sample of each period
* History of any significant cardiovascular disease
* Acute disease that generates significant physiological changes from the time of selection until the end of the study
* HIV, Hepatitis B and/or C positive
* Donation or loss of a significant volume (more than 100 mL) of blood or plasma or platelets during the 3 months prior to the start of the study
* Subjects who have participated in any type of clinical study during the 3 months prior to the start of the study
* History of any gastrointestinal surgery that could affect drug absorption
* Presence of fainting history or fear to blood collection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-02-27 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Total Duloxetine: area under the plasma concentration-time curve from 0 to 72 hours (AUC0-72) ] | From tablet intake and up to 72 hours after tablet intake
  17 samples up to 72 hours will be taken after the administration in each period.
Total Duloxetine: area under the plasma concentration-time curve from 0 to time t (AUC0-t) | From tablet intake and up to 72 hours after tablet intake
  17 samples up to 72 hours will be taken after the administration in each period.
Total Duloxetine: Maximum plasma concentration (Cmax) | From tablet intake and up to 72 hours after tablet intake
  17 samples up to 72 hours will be taken after the administration in each period.
Total Duloxetine: Time to achieve maximum plasma concentration (tmax) | Time Frame: From tablet intake and up to 72 hours after tablet intake
  17 samples up to 72 hours will be taken after the administration in each period.

CONTACTS AND LOCATIONS:
Locations (1):
- Innolab, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No